CLINICAL TRIAL: NCT01064427
Title: Factors Correlated With Fatigue in Breast Cancer Patients Before, During and After Adjuvant Chemotherapy
Brief Title: Factors Correlated With Fatigue in Breast Cancer
Acronym: FATSEIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Francis Guillemin, PU-PH, Inserm CIC-EC CIE6, CHU Nancy
Other Study IDs: 08-FATQV
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Newly Diagnosed Breast Cancer; Surgery Programmed
Keywords: breast cancer; fatigue; adjuvant chemotherapy; quality of life
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chemotherapy group: Breast cancer patients treated by adjuvant chemotherapy after their surgery. The time points of data collection are before the start of the first, second, fourth and sixth cycle of chemotherapy. If patients are treated by radiotherapy after the chemotherapy, there are 2 measurements points pre- and post radiotherapy.The others measurement points are at 12,18 and 24 months after surgery.
- No chemotherapy group: Breast cancer patients no treated by adjuvant chemotherapy after their surgery. For patients treated by radiotherapy after surgery, there are 2 measurement points pre- and post radiotherapy. The others measurement points are at 4,6,7,8,12,18 and 24 months after surgery.

SUMMARY:
The aim of this study is to identify the determinants of cancer-related fatigue, and the long-term effect of the different adjuvants treatments will be explored. A prospective longitudinal study in women diagnosed for the first time with stage I-III breast cancer and who have undergone surgery, has been designed to meet the study aims.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older
* newly diagnosed with stage I-IIIA breast adenocarcinoma
* have undergone surgery
* WHO performance status score equal or lower than 2
* able to provide informed consent
* speak French and able to complete self-report questionnaires

Exclusion Criteria:

* pregnancy
* bilateral breast cancer
* metastatic breast cancer
* patients who received neoadjuvant chemotherapy
* known psychiatric disease or dementia
* no previous history of cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment began in September 2008 and is planned over a 24-month period. Participants with breast cancer are recruited from three French cancer centers, the Alexis Vautrin anti-cancer center of Vandoeuvre-les-Nancy, the Georges-François Leclerc anti-cancer center of Dijon and the Paul Strauss anti-cancer center of Strasbourg, France. Participation to study is proposed to all women with newly diagnosed breast cancer the day preceeding surgery.Included patients are asked to complete the questionnaires several times.
Sampling Method: Probability Sample
Enrollment: 557 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The Multidimensional Fatigue Inventory (MFI-20) questionnaire is used to assess patient's fatigue. | Breast cancer patients complete the questionnaires before surgery and at several times depending on their adjuvant treatment

SECONDARY OUTCOMES:
Questionnaires regarding personality traits (LOT "Life Orientation Test" and the trait-version of the STAI "State Trait Anxiety instrument"), Quality of life questionnaire(EORTC QLQ-C30), and the state-version of the STAI will be also completed. | For the LOT and the trait-version of the STAI: only before the surgery, for the QLQ-C30: before surgery and several times during adjuvant treatment and for the state-version of the STAI: several times during adjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guillemin Francis, PU-PH, Principal Investigator — Inserm, CIC-EC CIE6, Nancy; CHU Nancy; Conroy Thierry, PU-PH, Principal Investigator — Centre Alexis Vautrin, Department of Medical Oncology, Vandoeuvre-les-Nancy, France
Locations (3):
- France (3):
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy, Meurthe et Moselle
  - Centre Georges François Leclerc, Dijon
  - Centre Paul Strauss, Strasbourg

REFERENCES:
- [Derived] Rotonda C, Guillemin F, Bonnetain F, Conroy T. Factors correlated with fatigue in breast cancer patients before, during and after adjuvant chemotherapy: the FATSEIN study. Contemp Clin Trials. 2011 Mar;32(2):244-9. doi: 10.1016/j.cct.2010.11.007. Epub 2010 Nov 13. PMID 21078419